CLINICAL TRIAL: NCT03825003
Title: Comparison of Joint Mobility Levels and Performance in Young Male Basketball Players and Sedentary Peers
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Begum Kara Kaya, Principal Investigator, Biruni University
Other Study IDs: 1
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2019-01

CONDITIONS: Hypermobility, Joint
Keywords: Basketball; Sedentary; Joint Mobility; Performance
MeSH Terms: conditions — Joint Instability; Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Basketball Players: Outcome assessments were done.
- Sedentary Peers: Outcome assessments were done.

SUMMARY:
The aim of our study was to determine the joint mobility levels and its effects on performance in male basketball players and their sedentary peers aged 16-22 years.

According to the studies on the effect of hypermobility on the performance; The young athletes who played tennis had lower equilibrium results than those without hypermobility. Although there is not any study that investigate its effects in basketball, there are studies for tennis and volleyball in literature.

ELIGIBILITY:
Inclusion Criteria:

For Players:

* Being a healthy male between the ages of 16-22,
* Playing basketball for at least 1 year,
* Body Mass Index <30,
* Volunteer to participate in research.

For Sedentary Peers:

* Being a healthy male between the ages of 16-22,
* International Physical Activity Questionnaire Short Form score <600 MET-min/week,
* Body Mass Index <30,
* Volunteer to participate in research.

Exclusion Criteria:

* To have a musculoskeletal problem which prevents the person from exercising,
* Having a cardiovascular system disorder that limits exercise capacity
* Neurological disorder or cognitive dysfunction
* Smoking

Ages: 16 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: The e-picos website was used to calculate the sample size. We used correlation coefficient (r = 0.505) from Acar et al's study in tennis players according to flamingo test results. When 90% power for each group is determined as α = 0.05, sample size is determined as 37. Considering the possibility of drop out by 10 percent, the sample size was determined as 41. 41 basketball players and 41 sedentary peers were included in the study.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Beighton Score | 1 day
  Beighton score is used to assess the levels of joint mobility in people. In this scoring, the lowest score is 0 and the highest score is 9. A total score of 4 and above is considered as joint hypermobility.
Y-Balance Test | 1 day
  Y balance test is used to evaluate dynamic balance in individuals. In the test setup, 3 pieces of tape measure are adhered to the floor in an angle of 120 degrees. At the intersection of 3 tapes, the subject is asked to stand on one foot and extend with the other foot in 3 directions, anterior, posteromedial and posterolateral. Test is repeated 3 times for each directions and the average score is recorded in cm. Higher score shows better performance.
Flamingo Balance Test | 1 day
  Flamingo ebalance test is used to evaluate static balance in individuals. The aim is to be able to balance successfully on the dominant barefoot. The subject is asked to step on the wooden wedge (50x4x3 cms) with the foot. He is asked to bend other foot to the back and to hold his foot with the same hand. Till maintaning the balance, subject holds the arm of tester. After he leaves the arm, test begins. The subject is asked to keep balance within 1 minute. The stopwatch is started as soon as the person leaves the arm of the tester. The stopwatch is stopped when the subject leaves each leg or any part of the body touches the ground. Any attemptation which maintain the balance during 1 minute is considered as score. Higher scores show better performance.
Vertical Jump Test | 1 day
  The vertical jump test is used to measure bounce strength and jump height. To perform the test, a special setup or a measurement system marked on the wall, chalk are required. The subject is asked to touch the highest point that he can reach out by extending his arm. This is called stopping height. It is important to note that the feet of the subject must be completely in contact with the ground. Then the subject is asked to reach the highest point by jumping. The difference between the height reached by the stop and the height reached by the jump give the score of test. The subject is asked to jump 3 times and the average score is recorded. Highest score shows better performance.
T Drill Test | 1 day
  T Drill test was used to assess agility and speed. 3 funnels are placed in line with a distance of 4.57 meters between them. Taking the starting point from the middle of the funnels (in the form of the letter T), it comprises a 9.14 meter forward fast run, 4.57 meter side step to the right, 9.14 meter side step to the right, 4.57 meter side step to the right and 9.14 meter backward to the right.The subject performs the test for three times. The average of the scores are recorded in seconds. Lower scores show better performance.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire-Short Form | 1 day
  International Physical Activity Questionnaire Short Form(IPAQ-SF) scales the types of intensity of physical activity and sitting time that people do as part of their daily lives. The short form records the physical activity of 3 different intensity levels: 1) vigorous-intensity activity such as aerobics (8.0 MET), 2) moderate-intensity activity such as leisure cycling (4.0 MET), 3) walking (3.3 MET). The IPAQ-SF questions activities for last 7 days with 7 items. In the scoring total estimate physical activity in MET-min/week and time spent while sitting are calculated ( Ex. 4.0 METx activity dayx activity duration (in minutes) equals moderate-intensity activity total MET score).According to scores subjects are categorized as inactive (achieving <600 MET-min/week), minimally active (achieving a minimum of at least 600 MET-min/week and <3000 MET-min/week), active (>3000 MET-min/week).

CONTACTS AND LOCATIONS:
Overall Officials: Begüm Kara Kaya, MSc, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No